CLINICAL TRIAL: NCT00791245
Title: A Post Market Study of Articular Cartilage Defects of the Knee Treated Wtih DeNovo NT, Natural Tissue Graft
Brief Title: Post Market Study of DeNovo NT, Natural Tissue Graft
Status: Completed | Type: Observational
Sponsor: Zimmer Orthobiologics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ISTO - DeNovo NT 03-07-02
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Last update posted 2014-08-11 (Estimated); Status verified 2014-08

CONDITIONS: Cartilage Repair
Keywords: ISTO Technologies, Inc; cartilage repair; arthroscopy; 361 HCT/P; human tissue; biologic; knee

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- 1: DeNovo NT
  Interventions: Biological: Particulated Juvenile Cartilage Allograft

INTERVENTIONS:
Biological: Particulated Juvenile Cartilage Allograft — Particulated Juvenile Cartilage Allograft

SUMMARY:
The purpose of this post market study is to evaluate surgical implantation technique and the quality of repair of the cartilage defect with particulated juvenile cartilage in the human knee joint.

DETAILED DESCRIPTION:
The intent of this post market study is to assess the clinical outcomes of DeNovo NT, a particulated juvenile cartilage tissue for the treatment of one or two contained lesion(s) equal to an ICRS Grade 3a, 3b, 3c, 3d of the femoral condyle or trochlear groove and OCD lesions (Grade 4a) with healed bone base, which is non sclerotic and no loss of bone greater thank 6mm measured from the surrounding subchondral plate.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary signature of the IRB approved Informed Consent
* Male or female subjects between the ages of 18 to 55 years
* If female:

  * Actively practicing a contraception method, or
  * Practicing abstinence, or
  * Surgically sterilized, or
  * Postmenopausal
* Pretreatment arthroscopic confirmation indicating one or two contained lesion(s) are equal to an ICRS Grade 3a, 3b, 3c, 3d of the femoral condyle or trochlear groove and OCD lesions (Grade 4a) with healed bone base, which is non sclerotic and no loss of bone greater than 6mm measured from the surrounding subchondral plate,
* Has peripheral cartilage debridement to healthy cartilage that results in a lesion(s) with an area of greater than or equal to 1 cm squared and less than or equal to 5 cm squared,
* PCL, LCL and MCL in the affected knee are stable and the ACL is stable or can be stabilized as a concomitant procedure,
* Ipsilateral knee compartment has intact menisci (or requires partial meniscectomy resulting in stable menisci),
* The contralateral knee is asymptomatic, stable and fully functional,
* Must be physically and mentally willing and able to comply with post-operative rehabilitation and routinely schedule clinical and radiographic visits through 24 months.

Exclusion Criteria:

* Clinical and/or radiographic disease diagnosis of the indexed affected joint that includes:

  * Osteoarthritis or avascular necrosis,
  * Rheumatoid arthritis, or history of septic or reactive arthritis,
  * Gout or a history of gout or pseudogout in the affected knee,
  * Osteochondritis dissecans of the knee with significant bone loss (greater than 6mm deep from the subchondral plate),
  * Associated damage to the underlying subchondral bone requiring an osteochondral graft,
* History of secondary arthropathies (i.e. sickle cell disease, hemochromatosis, or autoimmune disease),
* Uncontrolled diabetes,
* Displays a high surgical risk due to unstable cardiac and/or pulmonary disease,
* Has HIV or other immunodeficient state including subjects on immunosuppressant therapies, or has significant illness (metastasis of any type) that decreases the probability of survival to the 2 year endpoint,
* Is at substantial risk for the need of organ transplantation, such as renal insufficiency,
* Is pregnant or breast-feeding,
* Body Mass Index >35 (BMI=kg/m2),
* Has bipolar articular cartilage involvement or kissing lesions of the ipsilateral compartment, described as tibial or patellar lesions in the same compartment with greater than ICRS Grade 2 chondrosis,
* Is participating concurrently in another clinical trial, or has participated ina clinical trial within 30 days of surgery,
* Is receiving prescription pain medication other than NSAIDs or acetaminophen for conditions unrelated to the index knee condition, chronic use of anticoagulants, or taking corticosteroids,
* Has a neuromuscular, neurosensory, or musculoskeletal deficiency that limits the ability to perform objective functional assessment of either knee,
* Active joint infection,
* Prior total meniscectomy of either knee,
* Radiographically has >5 degrees of malalignment as measured from the hip, knee and ankle mechanical axis,
* Has received, within the past three months intra-articular hyaluronic acid therapy or cortisone injections in the index knee,
* Prior realignment surgery in the affected knee within the past 6 months,
* Failed microfracture treatment performed less than 12-months before baseline,
* Is receiving workman's compensation or currently involved in litigation relating to the index knee,
* Has history of alcoholism, medication or intravenous drug abuse, psychosis, is a prisoner, has a personality disorder(s), poor motivation, emotional or intellectual issues that would likely make the subject unreliable for the study, or any combination of variables in the investigator's judgement that should exclude a potential subject,
* Had or have an aneurysm clip implanted, intraocular foreign bodies (commonly seen in welders), subcutaneous metal shards (found in sheet metal workers), or some shrapnel; additionally no cardiac pacemaker, defibrillator, implanted neurostimulator (TENS implants), some prosthetic heart valve (especially mitral valve), cochlear implant or other hearing aid, or has a tendency of claustrophobia. Have tattoos that may contain iron-based dyes.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Clinical population
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2006-01; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
KOOS | Preoperatively, postoperatively at 10 Days, 3, 6, 12, 18 & 24 Months

SECONDARY OUTCOMES:
IKDC Subjective Knee Evaluation | Preopertively, postoperatively at 10 Days, 3, 6, 12, 18, & 24 Months

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Midwest Orthopaedics at Rush, Chicago, Illinois
  - OrthoIndy, Indianapolis, Indiana
  - New Mexico Orthopaedic Association, PC, Albuquerque, New Mexico